CLINICAL TRIAL: NCT00159081
Title: One Year Maintenance Treatment With Low Dose Haloperidol vs. Risperidone in First-Episode Schizophrenia
Brief Title: One Year Drug Treatment in First-Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Network On Schizophrenia (Network); Janssen-Cilag Ltd. (Industry); University of Bonn (Other); Humboldt-Universität zu Berlin (Other); University of München (Other); University of Göttingen (Other); University of Cologne (Other); Mainz University (Other); University Hospital Tuebingen (Other); Universität Duisburg-Essen (Other); University of Mannheim (Other); University of Jena (Other); Martin-Luther-Universität Halle-Wittenberg (Other); RWTH Aachen University (Other); University of Wuerzburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01GI 9932 - P 2.2.2.1 / 1
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; first episode; long-term treatment; typical vs. atypical neuroleptics
MeSH Terms: conditions — Schizophrenia | interventions — Haloperidol; Risperidone; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Maintenance antipsychotic treatment with risperidone
  Interventions: Drug: Haloperidol, Risperidone (drug)
- 2 (Active Comparator): Maintenance antipsychotic treatment with haloperidol in low-dose
  Interventions: Drug: Haloperidol, Risperidone (drug)

INTERVENTIONS:
Drug: Haloperidol, Risperidone (drug) — targeted dose of 2-4 mg/day over 1 year

SUMMARY:
Prospective, randomized, double-blind, multi-center study on 1 year course and treatment outcome under low-dose typical (haloperidol) vs. atypical neuroleptics (risperidone) in first-episode schizophrenia.

DETAILED DESCRIPTION:
The objective of this multi-center study is to optimize the long-term treatment of patients with first episode schizophrenia. This investigation should contribute to the issue of effective relapse prevention in first-episode patients. 1-year maintenance neuroleptic treatment is done with low dose haloperidol or risperidone (target dose 2-4 mg/die).

ELIGIBILITY:
Inclusion Criteria:

* After the acute treatment of the first-episode in schizophrenia (according ICD-10 F20)
* Age between 18 and 55
* Informed consent

Exclusion Criteria:

* Residence outside of the catchment area
* Legal reasons
* Insufficient knowledge of the German language
* Substance abuse or addiction
* Pregnancy
* Serious physical illness
* Organic brain disease
* Contraindication to neuroleptic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2000-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
relapse rate | 1 year

SECONDARY OUTCOMES:
course in psychopathology | 1 year
social and cognitive functioning | 1 year
side-effects | 1 year
drop-out | 1 year
quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Gaebel, Professor, Study Chair — Department of Psychiatry and Psychotherapy, University of Duesseldorf
Locations (1):
- Department of Psychiatry and Psychotherapy at the Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Gaebel W, Moller HJ, Buchkremer G, Ohmann C, Riesbeck M, Wolwer W, Von Wilmsdorff M, Bottlender R, Klingberg S. Pharmacological long-term treatment strategies in first episode schizophrenia--study design and preliminary results of an ongoing RCT within the German Research Network on Schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2004 Apr;254(2):129-40. doi: 10.1007/s00406-004-0509-y. PMID 15146342
- [Result] Gaebel W, Riesbeck M, Wolwer W, Klimke A, Eickhoff M, von Wilmsdorff M, Jockers-Scherubl MC, Kuhn KU, Lemke M, Bechdolf A, Bender S, Degner D, Schlosser R, Schmidt LG, Schmitt A, Jager M, Buchkremer G, Falkai P, Klingberg S, Kopcke W, Maier W, Hafner H, Ohmann C, Salize HJ, Schneider F, Moller HJ; German Study Group on First-Episode Schizophrenia. Maintenance treatment with risperidone or low-dose haloperidol in first-episode schizophrenia: 1-year results of a randomized controlled trial within the German Research Network on Schizophrenia. J Clin Psychiatry. 2007 Nov;68(11):1763-74. doi: 10.4088/jcp.v68n1116. PMID 18052570
- See also: Click here for more information about this study: One year maintenance treatment with low dose Haloperidol vs. Risperidone in first-episode schizophrenia — http://www.kompetenznetz-schizophrenie.de